CLINICAL TRIAL: NCT07004881
Title: Comparison Between the Effects of Mulligan and Maitland Mobilization on Patellofemoral Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/74
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-08

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: It is a single blinded Randomized Controlled Trial, in which the data assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization with Movement (Active Comparator): Mulligan Mobilization with Movement This group will receive two techniques of mulligan i.e. Medial Patellar Glide relative to femoral trochlea and other is tibial internal rotation relative to femoral condyles.
  Both the techniques are repeated 10 times with total 3 sets. 3 sessions are performed in a week on alternate days. Total duration of interventions is 2 weeks.
  After mobilization, following exercises are to be performed all in 3 sets of 7 repetitions:
  1. Side-lying hip abduction
  2. Clamshell exercises
  3. Quadriceps setting exercise
  4. Vastus Medialis Oblique strengthening
  5. Mini squats
  6. Hamstring stretch
  7. Iliotibial band stretch
  Interventions: Procedure: Group A (Active Comparator) Mulligan's Mobilization With Movement (MWM)
- Maitland Mobilization (Experimental): Maitland Mobilization This group recieves 4 patellar mobilization tehniques given by Maitland. For all the mobilizations the patient is positioned either in supine or sitting with 30-0 degree knee flexion or full knee extension.
  The therapist holds patella between his/her thumb and index finger and glides it cranially (Superior Patellar glide), caudally (Inferior Patellar Glide) and medially (Medial Patellar Glide).
  The fourth one i.e. Patellofemoral Distraction is given by grasping the patella between two fingers and lifting it above/away from underlying femoral trochlea. All 4 of these techniques are repeated 10 times with total 3 sets. 3 sessions are performed in a week on alternate days.
  Total duration of interventions is 2 weeks.
  After mobilization; 3 sets of 7 repetitions:
  1. Side-lying hip abduction
  2. Clamshell exercises
  3. Quadriceps setting exercise
  4. Vastus Medialis Oblique strengthening
  5. Mini squats
  6. Hamstring stretch
  7. Iliotibial band stretch
  Interventions: Procedure: Group B(Experimental) Maitland's Patellar Mobilizations

INTERVENTIONS:
Procedure: Group A (Active Comparator) Mulligan's Mobilization With Movement (MWM) — This group will receive two techniques of mulligan i.e. Medial Patellar Glide relative to femoral trochlea and other is tibial internal rotation relative to femoral condyles.In Medial Patellar Glide; patient is positioned supine with 40 degree knee flexion. Stabilizing hand of therapist stabilizes the posterior aspect of tibia and fibula and with mobilizing hand, the therapist gently glides the patella medially. With that, the patient is asked to actively flex and then extend the knee.
  In the tibial internal rotation technique; similarly the patient is positioned supine with 40 degree knee flexion. Stabilizing hand of therapist stabilizes t
  After mobilization; following exercises are to be performed all in 3 sets of 7 repetitions:
  1. Side-lying hip abduction
  2. Clamshell exercises
  3. Quadriceps setting exercise
  4. Vastus Medialis Oblique strengthening
  5. Mini squats
  6. Hamstring stretch
  7. Iliotibial band stretch
  Arms: Mulligan Mobilization with Movement
Procedure: Group B(Experimental) Maitland's Patellar Mobilizations — For all the mobilizations the patient is positioned either in supine or sitting with 30-0 degree knee flexion or full knee extension. The therapist holds patella between his/her thumb and index finger and glides it cranially (Superior Patellar glide), caudally (Inferior Patellar Glide) and medially (Medial Patellar Glide). The fourth one i.e. Patellofemoral Distraction is given by grasping the patella between two fingers and lifting it above/away from underlying femoral trochlea. All 4 of these techniques are repeated 10 times with total 3 sets. 3 sessions are performed in a week on alternate days. Total duration of interventions is 2 weeks.
  Both groups receive similar exercises therapy following mobilizations.
  Arms: Maitland Mobilization

SUMMARY:
This study is a randomised control trial and the purpose of this study is to investigate and compare the "Effects of Maitland mobilizations and Mulligan Mobilization With Movement (MWM) in patients with Patellofemoral Pain Syndrome

DETAILED DESCRIPTION:
This study is a randomised control trial just used to investigate and compare the effects of maitland mobilizations and Mulligan's Mobilization With Movement ; with respect to:

1. Pain
2. Range of motion and
3. Function in patients with Patellofemoral pain syndrome All males and females with ages of 18 to 40 years having the Patellofemoral pain syndrome can be included in this study.

A total number of 40 participants are equally and randomly divided into two groups i.e. group A and group B. Group A recieves the Mulligan Mobilization With Movement (MWM) and group B receives the Maitland's Patellar mobilizations.

Outcomes are recorded at 0 weeks and at end of 2 weeks. Outcome measure used for pain is Numeric Pain Rating Scale (NPRS), for knee ROM is goniometery and for knee function is Lower Extremity Function Scale (LEFS).

Pre and post intervention reading of all 3 measures will then be compared and data will be analysed

ELIGIBILITY:
Inclusion Criteria:

* Referred patients from rehabilitation, orthopedic and rheumatology department
* Both males and females of age 18-40 years
* Having pain from at least 2 months.
* Pain score ≥ 3 on NPRS.
* Pain on palpation of medial or lateral Patellar facet. (12, 13)
* Retro patellar pain in at least two of the following activities:
* Ascending , descending stairs
* Hopping / jumping
* prolonged sitting with flexed knees
* kneeling and squatting
* Patellar tilt test

  * EXCLUSION CRIETERIA:
* Positive tests/findings on physical examination for knee menisci, ligaments and bursa.
* Chondromalacia patellae
* Individuals with Instability of tibiofemoral joint
* lower extremity surgery
* Rheumatoid arthritis, other connective tissue disorders and congenital deformities.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Patellofemoral Pain | 2 weeks
  It will be measured using numeric pain rating scale (NPRS). Subjects select a number ranging from 0-10 according to their intensity of pain where '0' indicates no pain while '10' indicates worst pain experienced.
Range of Motion | Variable will be assessed at before and after treatment for the total interval of 2 weeks.
  Universal goniometer is used to measure knee flexion and extension ranges. Patient is positioned in supine with the knee straight and foot flat on the table. Therapist stabilizes the femur with one hand. Axis of goniometer is aligned with the lateral epicondyle of the femur, stationary arm is kept parallel to the femur and moving arm is aligned with long axis of tibia. The patient is then asked to flex and extend the knee to maximum range without pain, subsequently aligning moving arm of goniometer with new position of tibia. Angle of flexion/extension are then recorded from the goniometer and documented.
Lower Extremity Function | Variable will be assessed at before and after treatment for the total interval of 2 weeks.
  It is measured using Lower Extremity Function Scale (LEFS). The LEFS is a questionnaire used to assess an individual's ability to perform daily activities and functional tasks related to the lower extremities (hips, knees, ankles, and feet). It comprises of total 20 questions and patients rate their ability to perform each activity on a scale from 0 (unable to perform) to 4 (able to perform without difficulty). The total score ranges from 0 to 80, with higher scores indicating better functional ability. The total sore before and after interventions of both groups is calculated and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan